CLINICAL TRIAL: NCT06935162
Title: Teclistamab for Previously Treated Light-chain Amyloidosis Patients, a Phase II Study
Brief Title: Teclistamab in Previously Treated AL Amyloidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jian Li, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tec-001
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Focal Adhesion Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teclistamab (Experimental): Teclistamab will be administered via a subcutaneous injection
  Interventions: Drug: Teclistamab (Tec)

INTERVENTIONS:
Drug: Teclistamab (Tec) — Teclistamab will be administered via a subcutaneous injection

SUMMARY:
This is a phase II study in patients with previously treated immunoglobulin light-chain (AL) Amyloidosis to evaluate the efficacy and safety of teclistamab

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed AL amyloidosis
* Patients must have received at least one line of treatment, including daratumumab and bortezomib
* Relapse from previous treatment, or less than partial response after two cycles of treatment/less than very good partial response after three cycles of treatment
* dFLC > 50mg/L

Exclusion Criteria:

* Previous anti-BCMA targeted therapy
* Co-morbidity of uncontrolled infection
* Co-morbidity of other active malignancy
* Co-diagnosis of multiple myeloma or waldenstrom macroglobulinemia
* Co-morbidity of grade 2 Mobitz II or grade 3 atrioventricular block (expect for those with implanted pacemaker)
* Co-morbidity of sustained or recurrent nonsustained ventricular tachycardia
* Seropositive for human immunodeficiency virus
* Hepatitis B virus (HBV)-DNA > 1000 copies/mL
* Seropositive for hepatitis C (except in the setting of a sustained virologic response)
* Neutrophil <1×10E9/L, hemoglobin < 8g/dL, or platelet < 75×10E9/L.
* Severely compromised hepatic or renal function: alanine transaminase (ALT) or aspertate aminotransferase (AST) > 5 × upper limit of normal (ULN), total bilirubin > 2 × ULN, eGFR < 20 mL/min, or receiving renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematologic complete response (CR) at 3 months after treatment initiation | at 3 months after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No